CLINICAL TRIAL: NCT03294434
Title: Predicting Sites of Tumour Progression in the Invasive Margin of Glioblastomas (PRaM-GBM Study)
Acronym: PRaM-GBM
Status: Completed | Type: Observational
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Cancer Research UK (Other); Experimental Cancer Medicine Centres (Other)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, CCTU-Cancer Theme, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: PRaM-GBM
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients that consent to participate in the optional PET sub-study will consent to the collection of additional tissue biopsies to be taken at the time of their standard of care surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High Grade Glioma: Diffusion tensor Imaging (DTI-MRI) scan to be performed pre-operatively and pre-radiotherapy
  Interventions: Other: Diffusion tensor Imaging (DTI)

INTERVENTIONS:
Other: Diffusion tensor Imaging (DTI) — Diffusion tensor Imaging (DTI) is a technique sensitive to the ordered diffusion of water along white matter tracts and can detect subtle disruption. A diffusion tensor signature method was developed that splits the tensor information into isotropic and anisotropic diffusion components. This can differentiate regions of pure tumour from invaded white matter.

SUMMARY:
Brain tumours are the leading cause of cancer deaths in children, men under the age of 45 and women under the age of 25. Glioblastoma is the most common and most malignant primary tumour. The predominant treatment is surgical removal of the tumour followed by radiotherapy. Sadly the majority of patients given this treatment develop recurrent and progressive disease.

Better understanding of the invasive margin might improve outcomes by facilitating more complete surgical resection beyond the traditional contrast enhancing margins. Diffusion tensor MRI (DTI) is an imaging technique which may be able to predict the site of tumour recurrence. DTI has previously been shown to identify regions, which have been confirmed with biopsies, to be areas of invasive tumours and are present before progression is seen with an MRI.

The primary aim of this study is to qualify an imaging biomarker that can be applied at initial presentation, that can accurately predict the site of where glioblastomas will progress after treatment and allow personalisation of both radiotherapy and surgical targets.

DETAILED DESCRIPTION:
This is a multicentre, prospective longitudinal observational cohort study in patients with high grade glioma, who have surgery planned to remove >90% of the tumour, and subsequent radical radiotherapy with concomitant tomozolomide. The purpose of this study is to establish a model using DTI that can accurately predict the site of where glioblastomas will progress after treatment. This study aims to validate the use of DTI as a biomarker across multiple centres to develop analysis methods that could be used in the future to personalise radiotherapy treatment volumes, and potentially surgical targets.

Patients will be given a DTI-MRI both prior to the operation and prior to radiotherapy. Clinical MRIs will take place according to standard guidelines. Whilst the study is open patients will participate in the study until death. Once a total of 70 patients from the first 90 have shown true progression patients will participate in the study for a minimum of 6 months from the beginning of radiotherapy.

This study will be conducted in 6-10 NHS centres, where 120 patients will be recruited, patients who are withdrawn will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Assessed by a neuroscience MDT to have a high grade glioma on imaging, OR if in the opinion of the CI, with guidance from the local PI that all relevant and appropriate members of a multidisciplinary team agree a high grade glioma diagnosis;
* Considered suitable for radical radiotherapy (60 Gy) with concomitant chemotherapy (Stupp Regime);
* WHO PS 0 or 1 (see Appendix 3);
* Age ≥16;
* Patient suitable for tumour resection where the treating neurosurgeon feels that >90% of the enhancing tumour will be resected;

Exclusion Criteria:

* Patients who are participating in trials involving investigational treatments
* Patients who are unsuitable for a contrast-enhanced MRI will be excluded. Such clinical problems include, but are not limited to:
* MR unsafe metallic implants;
* Claustrophobia;
* Allergy to gadolinium contrast agent;
* History of severe renal impairment.
* Patients unable to provide written informed consent
* PET sub-study only: Pregnant women

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients aged 16 and over with newly diagnosed glioblastomas
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Site of glioblastoma true progression correctly predicted by DTI scan | 18 months
  Assess the diagnostic accuracy of DTI at pre-surgery or/and pre-radiotherapy as a biomarker to predict site of glioblastoma progression

SECONDARY OUTCOMES:
Accuracy of DTI as a biomarker | 18 months
  Explore difference of DTI performed pre-surgery and pre-radiotherapy to predict the site of glioblastoma progression
Perfusion imaging | 18 months
  Investigate dynamic susceptibility imaging to measure rCBV of the invasive margin to improve the accuracy of the DTI biomarker.
Time to progression | 18 months
  Investigate if pattern of invasion can predict time to progression
Extent of resection and volume of tumour that remains post-surgery by standard imaging and DTI | 18 months
  Determine the effect of resection on the invasive margin as determined by DTI
Radiotherapy dose according to DTI-defined invasive region | 18 months
  Retrospectively compare dose of radiotherapy using the DTI-defined invasive region receives with conventional radiotherapy plans

OTHER OUTCOMES:
Difference of area highlighted by amino-acid PET and DTI-MRI | 18 months
  Investigate the relationship between amino-acid PET, area of surgical resection and the area highlighted by DTI-MRI
Number of amino-acid PET only image guided biopsies taken from patients | 18 months
  Investigate the feasibility of taking image-guided biopsies from patients in the region outside of the area with increased amino-acid PET uptake
Site of glioblastoma true progression correctly predicted from pre-operative imaging by a region that is predicted by the DTI abnormality outside of the area of increased uptake to amino-acid on PET | 18 months
  Explore the extent of invasive disease (from DTI/perfusion) that is likely to be left following surgery by assessing potential resected tumour using amino acid PET

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Price, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No